CLINICAL TRIAL: NCT00545246
Title: A Phase I, Dose-Escalation Study of the Safety, Tolerability, and Pharmacokinetics of Intravenous Aflibercept in Combination With Intravenous Docetaxel Administered Every 3 Weeks in Patients With Advanced Solid Malignancies
Brief Title: A Phase I Study of Intravenous Aflibercept in Combination With Docetaxel in Japanese Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCD10091
Record Dates: First submitted 2007-10-16; First posted 2007-10-17 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Neoplasms
Keywords: VEGF Trap
MeSH Terms: conditions — Neoplasms | interventions — aflibercept; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- aflibercept + docetaxel (Experimental)
  Interventions: Drug: aflibercept (AVE0005); Drug: docetaxel

INTERVENTIONS:
Drug: aflibercept (AVE0005) — intravenous infusion
Drug: docetaxel — intravenous infusion

SUMMARY:
The primary objective of this study is to determine the dose of aflibercept to be further studied in combination with docetaxel in Japanese cancer patients.

The secondary objectives of this study are to assess the safety profile of aflibercept, to determine the pharmacokinetics of aflibercept, to make a preliminary assessment of antitumor effects.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed cancer patients without standard of care
* ECOG performance status 0 or 1
* Adequate organ and bone marrow function

Exclusion Criteria:

* Need for a major surgery or radiation therapy during the study
* History of hypersensitivity to docetaxel or polysorbate 80
* Treatment with chemotherapy, hormonal therapy, radiotherapy within 28 days
* Uncontrolled hypertension
* History of brain metastases
* Ascites requiring drainage
* Pregnancy or breastfeeding
* Patients who have previously been treated with aflibercept.

The investigator will evaluate whether there are other reasons why a patient may not participate.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-10; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) defined as grade 3 or higher National Cancer Institute - Common Terminology Criteria (NCI-CTC) toxicities | first 3-week cycle

SECONDARY OUTCOMES:
safety: physical examination, laboratory safety tests, adverse events | up to 60 days after last treatment
pharmacokinetic values | every 3-week cycle
objective response rate | every 3-week cycle

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (2):
- Japan (2):
  - Sanofi-Aventis Investigational Site Number 392002, Iruma-gun
  - Sanofi-Aventis Investigational Site Number 392001, Sunto-Gun

REFERENCES:
- [Derived] Sunakawa Y, Takahashi K, Kawaguchi O, Yamamoto N. Phase I study of aflibercept in combination with docetaxel in Japanese patients with advanced solid malignancies. Invest New Drugs. 2022 Oct;40(5):1032-1041. doi: 10.1007/s10637-022-01267-x. Epub 2022 Jun 30. PMID 35771301